CLINICAL TRIAL: NCT04835116
Title: Comparison of Post-Operative Analgesia With Peri Tract Local Anesthesia Infiltration and Oral Analgesia Versus Post-Operative Intravenous Analgesia After Percutaneous Nephrolithotomy.
Brief Title: Comparison of Post-Operative Analgesia After Percutaneous Nephrolithotomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Armed Forces Institute of Urology, Rawalpindi (Other)
Responsible Party: Principal Investigator, Musab Umair Khalid, Doctor, Armed Forces Institute of Urology, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFIU Rawalpindi
Record Dates: First submitted 2021-03-28; First posted 2021-04-08 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Pain; Postoperative Pain
Keywords: Local anesthesia, Percutaneous nephrolithotomy.
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Bupivacaine; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local Anesthesia (Other): Group A patients received peri tract local anaesthesia infiltration with 0.25% Bupivacaine.
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection. Paracetamol 650mg. Orphenadrine 50mg.; Drug: paracetamol 1000mg. Tramadol 50mg. Dimenhydrinate 50mg.
- Intravenous Analgesics (Other): Group B patients received postoperative intravenous analgesia.
  Interventions: Drug: Bupivacaine Hydrochloride 0.25% Injection. Paracetamol 650mg. Orphenadrine 50mg.; Drug: paracetamol 1000mg. Tramadol 50mg. Dimenhydrinate 50mg.

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.25% Injection. Paracetamol 650mg. Orphenadrine 50mg. — Group A patients were administered per-operative peri tract local anesthesia infiltration with 0.25% bupivacaine augmented by post-operative oral analgesia with a combination of Paracetamol 650 mg and Orphenadrine 50mg 6 hourly.
  Other Names: Local Anesthesia
Drug: paracetamol 1000mg. Tramadol 50mg. Dimenhydrinate 50mg. — Group B patients were only given post-operative intra-venous analgesia by Paracetamol 1gm intravenous 8 hourly augmented with a combination of Tramadol 50mg and Dimenhydrinate 50mg as and when required
  Other Names: Intravenous analgesic

SUMMARY:
The rationale of this study was to compare the efficacy of peri-tract bupivacaine infiltration with intravenous post-operative analgesia following PCNL in reference to the context with the previous studies so that we can adopt the better technique to curtail the post-operative pain.

DETAILED DESCRIPTION:
The rationale of this study was to compare the efficacy of peri-tract bupivacaine infiltration with intravenous postoperative analgesia following PCNL in reference to the context with the previous studies so that we can adopt the better technique to curtail the post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing PCNL
* age from 12-65 years
* normal renal functions
* no history of chronic pain
* ASA I, II & III
* Both genders

Exclusion Criteria:

* history of local anaesthesia allergy
* Redo PCNL
* Multiple punctures during PCNL
* Excessive intra-operative bleeding
* Diabetes mellitus
* Coagulopathy
* Mental disorder
* ASA IV & V
* Active urinary tract infection.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Comparison of Post-Operative Analgesia With Peri Tract Local Anesthesia Infiltration and Oral Analgesia Versus Post-Operative Intravenous Analgesia After Percutaneous Nephrolithotomy. | 6 months
  Efficacy of peri-tract infiltration of bupivacaine over standard oral analgesia in patients undergoing PCNL.
  Measurement: Postoperative pain Measurement tool: Visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Musab Umair, MBBS, Principal Investigator — Armed Forces Institute of Urology.
Locations (1):
- Armed Forces Institute of Urology., Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No